CLINICAL TRIAL: NCT01902134
Title: A Randomized, Double-blind, Placebo and Active-controlled, Parallel-group Study to Evaluate the Analgesic Efficacy and Safety of Dexketoprofen Trometamol and Tramadol Hydrochloride Oral Fixed Combination on Moderate to Severe Acute Pain After Elective Unilateral Total Hip Arthroplasty
Brief Title: Oral Treatment for Orthopaedic Post-operative Pain With Dexketoprofen Trometamol and Tramadol Hydrochloride
Acronym: DAVID-art
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Menarini Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DEX-TRA-05; 2012-004548-31 (EudraCT Number)
Record Dates: First submitted 2013-07-15; First posted 2013-07-18 (Estimated); Results first posted 2015-04-01 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2016-02

CONDITIONS: Acute Pain
Keywords: Moderate to severe acute pain; Postoperative pain; Hip arthroplasty; Analgesics; Dexketoprofen; Tramadol
MeSH Terms: conditions — Acute Pain; Pain, Postoperative | interventions — dexketoprofen trometamol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- DKP/TRAM followed by DKP/TRAM (Experimental): Dexketoprofen/Tramadol-single dose followed by Dexketoprofen/Tramadol-multiple doses
  Interventions: Drug: Dexketoprofen/Tramadol-single dose; Drug: Dexketoprofen/Tramadol-multiple doses
- DKP followed by DKP (Active Comparator): Dexketoprofen-single dose followed by Dexketoprofen-multiple doses
  Interventions: Drug: Dexketoprofen-single dose; Drug: Dexketoprofen-multiple doses
- TRAM followed by TRAM (Active Comparator): Tramadol-single dose followed by Tramadol-multiple doses
  Interventions: Drug: Tramadol-single dose; Drug: Tramadol-multiple doses
- Placebo followed by DKP/TRAM (Other): Placebo single dose followed by Dexketoprofen/Tramadol-multiple doses
  Interventions: Drug: Placebo; Drug: Dexketoprofen/Tramadol-multiple doses
- Placebo followed by DKP (Other): Placebo single dose followed by Dexketoprofen-multiple doses
  Interventions: Drug: Placebo; Drug: Dexketoprofen-multiple doses
- Placebo followed by TRAM (Other): Placebo single dose followed by Tramadol-multiple doses
  Interventions: Drug: Placebo; Drug: Tramadol-multiple doses

INTERVENTIONS:
Drug: Placebo — Placebo single oral dose (first 8 hours)
  Arms: Placebo followed by DKP; Placebo followed by DKP/TRAM; Placebo followed by TRAM
Drug: Tramadol-single dose — Tramadol single oral dose (first 8 hours)
  Arms: TRAM followed by TRAM
Drug: Dexketoprofen-single dose — Dexketoprofen single oral dose (first 8 hours)
  Arms: DKP followed by DKP
Drug: Dexketoprofen/Tramadol-single dose — Dexketoprofen/Tramadol oral single dose (first 8 hours)
  Arms: DKP/TRAM followed by DKP/TRAM
Drug: Tramadol-multiple doses — Tramadol multiple oral doses t.i.d. for 5 days (total 12 doses)
  Arms: Placebo followed by TRAM; TRAM followed by TRAM
Drug: Dexketoprofen-multiple doses — Dexketoprofen multiple oral doses t.i.d. for 5 days (total 12 doses)
  Arms: DKP followed by DKP; Placebo followed by DKP
Drug: Dexketoprofen/Tramadol-multiple doses — Dexketoprofen/Tramadol multiple oral doses t.i.d. for 5 days (total 12 doses)
  Arms: DKP/TRAM followed by DKP/TRAM; Placebo followed by DKP/TRAM

SUMMARY:
This study aims to evaluate the analgesic efficacy of single and repeated doses of fixed combination of dexketoprofen trometamol (DKP) and tramadol hydrochloride (TRAM) in comparison to the single agents (and placebo for the single dose phase only) Approximately 600 male and female patients presenting moderate to severe pain after an elective primary hip arthroplasty are eligible to be randomised provided that they experience moderate to severe pain on the day after surgery.

DETAILED DESCRIPTION:
In this clinical trial patients were randomized to the described 6 treatment arms, where each arm define the treatment to be received in the first single dose phase (lasting 8 hours after the 1st treatment intake) and in the subsequent multiple-dose phase (lasting from the second treatment intake up to the 8 hours after the last intake). Namely:

* DKP/TRAM followed by DKP/TRAM;
* DKP followed by DKP;
* TRAM followed by TRAM;
* placebo followed by DKP;
* placebo followed by TRAM;
* placebo followed by DKP/TRAM;

The analyses of endpoints pertinent to the single dose phase were performed combining all the 3 treatment arms including placebo into one group, which resulted in the following 4 analysis groups: DKP/TRAM, DEXKETOPROFEN, TRAMADOL, and Placebo.

The analysis of endpoints pertinent to the multiple dose phase were performed combining the treatment arms including the same active treatment, which resulted in the following 3 analysis groups: DKP/TRAM, DEXKETOPROFEN, and TRAMADOL.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 18 to 80 years. Females participating in the study must be either of non-childbearing potential, or willing to use a highly effective contraceptive method.
* Scheduled to undergo standard primary (first-time) one-sided total hip replacement surgery due to primary osteoarthritis.
* Patients experiencing pain at rest of at least moderate intensity the day after surgery.

Exclusion Criteria:

* Patients not suitable for study treatments and rescue medication (RM) or those for whom non-steroidal anti-inflammatory drugs (NSAIDs), opioids, acetyl salicylic acid, pyrazolones or pyrazolidines are contraindicated.
* Patients with clinically significant abnormalities in vital signs, safety laboratory tests and 12-lead ECG at screening.
* Patients with history of any illness or condition that might pose a risk to the patient or confound the efficacy and safety study results.
* Patients using and not suitable to withdraw analgesics other than those specified in the protocol.
* Patients using and not suitable for withdrawing any of the prohibited medication specified in the protocol.
* Pregnant and breastfeeding women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 641 (Actual)
Dates: Start 2013-04; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Moore, Professor, Study Chair — Pain Research & Nuffield Department of Anaesthetics - University of Oxford; Henry J McQuay, Professor, Study Chair — Balliol College Oxford
Locations (37):
- Czechia (5):
  - Fakultni nemocnice Brno, Brno
  - Urazova nemocnice v Brne, Brno
  - Nemocnice Jihlava, p.o., Jihlava
  - Oblastni nemocnice Kladno, Kladno
  - Oblastni nemocnice Mlada Boleslav a.s., Mladá Boleslav
- Klinikum Frankfurt Höchst GmbH, Frankfurt am Main, Germany
- Hungary (5):
  - Uzsoki Hospital, Department of Orthopaedics, Budapest
  - University of Debrecen, Debrecen
  - PTE KK Trauma Központ-Balesetsebészeti és Kézsebésze, Pécs
  - Fejér Megyei Szent György Kórház, Székesfehérvár
  - MÁV Kórház és Rendelőintézet, Ortopédiai osztály, Szolnok
- Latvia (4):
  - Liepaja Regional Hospital, Liepāja
  - Riga's 2nd Hospital, Riga
  - Hospital of Traumatology and Orthopaedics, Riga
  - Vidzemes Hospital, Valmiera
- Lithuania (4):
  - Kaunas Clinical Hospital, Kaunas
  - Hospital of Lithuanian University of Health Sciences Kaunas, Kaunas
  - Klaipedos Universitetine ligonine, Klaipėda
  - Respublikine Vilniaus universitetine ligonine, Vilnius
- Poland (6):
  - Uniwersytecki Szpital Klioniczny w Bialymstoku, Bialystok
  - Warminskie Centrum Ortopedyczne, Elblag
  - Wojewodzki Szpital Specjalistyczny, Lublin
  - Specjalistyczny Szpital im. E. Szczeklika, Tarnów
  - Urazowo - Ortopedycznej Wojewodzkiego Szpitala Specjalistycznego we Wrocławiu, Wroclaw
  - Medical University of Lodz, Lodz, Łódź Voivodeship
- Serbia (4):
  - Clinical Center of Serbia, Belgrade
  - Institute for orthopedic Surgery Banjica [Ortopedic Surgery, Belgrade
  - Clinical Center Kragujevac, Kragujevac
  - Clinic for Orthopedic Surgery and Trauma Bul. Dr Zorana Djindjica, Niš
- Spain (2):
  - Hospital L'Esperança. Parc de Salut Mar., Barcelona
  - Hospital Universitario Puerta del Mar, Cadiz
- Taiwan (2):
  - China Medical University Hospital [Orthopedic], Taichung
  - Kuang Tien General Hospital, Taichung
- Ukraine (4):
  - Cherkaska oblasna likarnia, Cherkasy
  - Instytut patologii khrebta ta suglobiv im. prof. M.I. Sytenka NAMN Ukraine, Kharkiv
  - Kyivska oblasna klinichna likarnia, Kyiv
  - Sevastopolska miska likarnia №9, Sevastopol

REFERENCES:
- [Result] McQuay HJ, Moore RA, Berta A, Gainutdinovs O, Fulesdi B, Porvaneckas N, Petronis S, Mitkovic M, Bucsi L, Samson L, Zegunis V, Ankin ML, Bertolotti M, Piza-Vallespir B, Cuadripani S, Contini MP, Nizzardo A. Randomized clinical trial of dexketoprofen/tramadol 25 mg/75 mg in moderate-to-severe pain after total hip arthroplasty. Br J Anaesth. 2016 Feb;116(2):269-76. doi: 10.1093/bja/aev457. PMID 26787797

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Followed by DKP: Placebo single dose followed by Dexketoprofen-multiple doses Placebo followed by DKP
Period: Overall Study
Arm/Group | DKP/TRAM Followed by DKP/TRAM | DKP Followed by DKP | TRAM Followed by TRAM | Placebo Followed by DKP/TRAM | Placebo Followed by DKP | Placebo Followed by TRAM
Started | 159 | 161 | 160 | 54 | 53 | 54
Single-dose Phase | 159 | 161 | 160 | 54 | 53 | 54
Multiple-dose Phase | 159 | 160 | 160 | 54 | 53 | 52
Completed | 151 | 150 | 145 | 52 | 46 | 45
Not Completed | 8 | 11 | 15 | 2 | 7 | 9
Not completed — Adverse Event | 3 | 1 | 2 | 1 | 1 | 3
Not completed — Lack of Efficacy | 0 | 0 | 2 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 4 | 8 | 9 | 1 | 5 | 4
Not completed — no compliance | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 1 | 2 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intention-to-treat (ITT) population (which includes all patients randomized).
Groups:
- Total: Total of all reporting groups
Arm/Group | DKP/TRAM Followed by DKP/TRAM | DKP Followed by DKP | TRAM Followed by TRAM | Placebo Followed by DKP/TRAM | Placebo Followed by DKP | Placebo Followed by TRAM | Total
Number analyzed (Participants) | 159 | 161 | 160 | 54 | 53 | 54 | 641
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (10.43) | 63.3 (9.01) | 61.3 (9.68) | 63.9 (9.0) | 61.0 (11.10) | 59.8 (11.30) | 61.9 (9.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 86 | 80 | 37 | 33 | 24 | 346
  Male | 73 | 75 | 80 | 17 | 20 | 30 | 295
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 0 | 2 | 3 | 0 | 0 | 2 | 7
  White | 159 | 159 | 157 | 54 | 53 | 52 | 634
Region of Enrollment [Number; unit: participants]
  Serbia | 15 | 18 | 14 | 5 | 5 | 5 | 62
  Taiwan | 0 | 2 | 3 | 0 | 0 | 2 | 7
  Czech Republic | 9 | 10 | 8 | 2 | 4 | 3 | 36
  Hungary | 49 | 57 | 54 | 17 | 16 | 11 | 204
  Spain | 1 | 0 | 1 | 0 | 0 | 0 | 2
  Poland | 10 | 8 | 8 | 2 | 2 | 3 | 33
  Ukraine | 15 | 13 | 13 | 6 | 6 | 3 | 56
  Lithuania | 22 | 19 | 21 | 6 | 5 | 11 | 84
  Germany | 1 | 1 | 2 | 0 | 0 | 0 | 4
  Latvia | 37 | 33 | 36 | 16 | 15 | 16 | 153
Weight [Mean (Standard Deviation); unit: kg] | 83.3 (15.37) | 81.4 (15.63) | 83.5 (17.25) | 82.4 (15.91) | 81.7 (13.77) | 82.1 (15.27) | 82.6 (15.80)
Height [Mean (Standard Deviation); unit: cm] | 168.8 (8.99) | 167.9 (9.14) | 169.1 (9.20) | 166.1 (8.47) | 168.0 (9.49) | 169.9 (7.94) | 168.5 (9.01)

OUTCOME MEASURES:

1. Primary Outcome: SPID8 (Sum of Pain Intensity Differences Over 8 Hours)
Description: Sum of Pain Intensity Differences calculated as the weighted sum of the PI-VAS differences over 8 hour period. PI-VAS corresponds to the pain intensity measured by a 0-100 visual analogue scale (0=no pain to 100=worst pain imaginable) which was measured at 0.5h, 1h, 1.5h, 2h, 3h, 4h, 6h, and 8h after the first dose. A higher value in SPID indicates greater pain relief.
  The analysis was performed combining all randomization arms including placebo into one group, which resulted in the following 4 analysis groups: DKP/TRAM, DEXKETOPROFEN, TRAMADOL, and Placebo.
Time Frame: over 8 hours after the first dose
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- DKP/TRAM: Drug: Dexketoprofen/Tramadol single oral dose (first 8 hours); Arm type: experimental; Dexketoprofen/Tramadol single oral dose (first 8 hours);
- DEXKETOPROFEN: Drug: Dexketoprofen single oral dose (first 8 hours); Arm type: active comparator; Dexketoprofen single oral dose (first 8 hours);
- TRAMADOL: Drug: Tramadol single oral dose (first 8 hours); Arm type: active comparator; Tramadol single oral dose (first 8 hours);
- PLACEBO: Drug: Placebo; Arm type: PLACEBO comparator; Placebo single oral dose (first 8 hours);
Arm/Group | DKP/TRAM | DEXKETOPROFEN | TRAMADOL | PLACEBO
Number analyzed (Participants) | 159 | 161 | 160 | 161
units on a scale | 246.9 (156.50) | 208.8 (154.69) | 204.6 (145.79) | 151.1 (158.51)

2. Secondary Outcome: SPID48 (Sum of Pain Intensity Differences Over First 48 Hours of the Multiple-dose Phase)
Description: Sum of Pain Intensity Differences calculated as the weighted sum of the PI-VAS differences over 48 hours of the multiple-dose phase.
  PI-VAS corresponds to the pain intensity measured by a 0-100 visual analogue scale (0=no pain to 100=worst pain imaginable) which was measured every two hours over the first 48 hours of the multiple-dose phase. A higher value in SPID indicates greater pain relief.
  The analysis was performed combining all randomization arms including the same active treatment, which resulted in the following 3 analysis groups: DKP/TRAM, DEXKETOPROFEN, and TRAMADOL.
Time Frame: over 48 hours of the multiple-dose phase
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- DKP/TRAM: Drug: Dexketoprofen/Tramadol multiple doses; Arm type: experimental; Dexketoprofen/Tramadol multiple oral doses t.i.d. for 5 days (a total of 12 doses)
- DEXKETOPROFEN: Drug: Dexketoprofen multiple doses; Arm type: active comparator; Dexketoprofen multiple oral doses t.i.d. for 5 days (a total of 12 doses)
- TRAMADOL: Drug: Tramadol multiple doses; Arm type: active comparator; Tramadol multiple oral doses t.i.d. for 5 days (a total of 12 doses)
Arm/Group | DKP/TRAM | DEXKETOPROFEN | TRAMADOL
Number analyzed (Participants) | 213 | 214 | 214
units on a scale | 1943.7 (1000.51) | 1677.5 (1070.91) | 1765.6 (963.49)

3. Secondary Outcome: Percentage of Responders According to PI-VAS (Pain Intensity - Visual Analogue Scale)
Description: Percentage of responders; response defined as achievement a mean pain intensity, PI-VAS < 40 mm (PI-VAS corresponds to the pain intensity measured by a 0-100 visual analogue scale, 0=no pain to 100=worst pain imaginable),over 48 hours of the multiple-dose phase.
  The analysis was performed combining all randomization arms including the same active treatment, which resulted in the following 3 analysis groups: DKP/TRAM, DEXKETOPROFEN, and TRAMADOL.
Time Frame: over 48 hours of the multiple-dose phase
Measure: Number; unit: percentage of participants
Arm/Group | DKP/TRAM | DEXKETOPROFEN | TRAMADOL
Number analyzed (Participants) | 213 | 214 | 214
percentage of participants | 90.1 | 76.6 | 82.2

4. Secondary Outcome: Percentage of Responders According to 50% Max TOTPAR (Total Pain Relief)
Description: Percentage of responders over 8 hours after first dose, according to the 50% maximum total pain relief rule: maximum TOTPAR calculated as the theoretical maximum weighted sum of PAR-VRS (Pain Relief - Verbal Rating Scale: pain relief 0=none, 4=complete) scores.
  The analysis was performed combining all randomization arms including placebo into one group, which resulted in the following 4 analysis groups: DKP/TRAM, DEXKETOPROFEN, TRAMADOL, and Placebo.
Time Frame: over 8 hours after the first dose
Measure: Number; unit: percentage of participants
Groups:
- PLACEBO: Drug: Placebo; Arm type: PLACEBO comparator; Placebo single oral dose during single dose phase (first 8 hours);
Arm/Group | DKP/TRAM | DEXKETOPROFEN | TRAMADOL | PLACEBO
Number analyzed (Participants) | 159 | 161 | 160 | 161
percentage of participants | 57.9 | 56.5 | 51.9 | 37.9

ADVERSE EVENTS:
Time Frame: Study duration for patients was up to 6 weeks.
Description: Analyzed for the Safety population (all randomized patients who received at least one dose of the study treatment). Includes adverse events emerging after at least one dose of active study treatment.
Arm/Group | DKP/TRAM Followed by DKP/TRAM | DKP Followed by DKP | TRAM Followed by TRAM | Placebo Followed by DKP/TRAM | Placebo Followed by DKP | Placebo Followed by TRAM
Serious Adverse Events (participants affected / at risk) | 2/159 | 3/161 | 1/160 | 1/54 | 0/53 | 0/54
Other Adverse Events (participants affected / at risk) | 15/159 | 18/161 | 24/160 | 9/54 | 2/53 | 5/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DKP/TRAM Followed by DKP/TRAM (N=159) | DKP Followed by DKP (N=161) | TRAM Followed by TRAM (N=160) | Placebo Followed by DKP/TRAM (N=54) | Placebo Followed by DKP (N=53) | Placebo Followed by TRAM (N=54)
Bone operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Heart valve replacement (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular graft (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device dislocation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Face oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac disorder (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periorbital oedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DKP/TRAM Followed by DKP/TRAM (N=159) | DKP Followed by DKP (N=161) | TRAM Followed by TRAM (N=160) | Placebo Followed by DKP/TRAM (N=54) | Placebo Followed by DKP (N=53) | Placebo Followed by TRAM (N=54)
Anaemia postoperative (Injury, poisoning and procedural complications) | 7 (7) | 6 (6) | 5 (5) | 3 (3) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 4 (4) | 9 (9) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 9 (10) | 11 (12) | 3 (3) | 2 (3) | 4 (5)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to submitting the results of this study for publication or presentation, the PI will allow the Sponsor at least 60 days to review and comment upon the publication manuscript. The Sponsor will provide any manuscript of the results of this study at least 60 days before publishing to the authors for a complete review.